CLINICAL TRIAL: NCT03432637
Title: Thoracoscopic Lobecotmy Under Spontaneous Ventilating Anesthesia or Intubated Anesthesia: A Prospective, Multicentre, Open-label, Randomized Control Trial
Brief Title: Clinical Trial of Thoracoscopic Lobecotmy Under Spontaneous Ventilating Anesthesia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Shenzhen People's Hospital (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, Jun Liu, Principal Investigator, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVA-NSCLC
Record Dates: First submitted 2018-01-31; First posted 2018-02-14 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Complications, Postoperative/Perioperative; video assisted thoracic surgery; non-intubated anaesthesia
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SV (Experimental): undergoing thoracoscopic lobectomy under spontaneous ventilation (SV)
  Interventions: Procedure: spontaneous ventilation
- SLV (Active Comparator): undergoing thoracoscopic lobectomy under intubated anesthesia with single-lung mechanical ventilation(SLV)
  Interventions: Procedure: intubated anesthesia with single-lung mechanical ventilation

INTERVENTIONS:
Procedure: spontaneous ventilation — thoracoscopic lobectomy under spontaneous ventilation
  Arms: SV
Procedure: intubated anesthesia with single-lung mechanical ventilation — undergoing thoracoscopic lobectomy under intubated anesthesia with single-lung mechanical ventilation
  Arms: SLV

SUMMARY:
With the development of video-assisted thoracoscopic surgery (VATS) techniques and technology for anesthesia control, non-intubated anesthesia with spontaneous ventilation has been widely applied in VATS. A prospective, multicentre, randomized controlled clinical study was applied in this study to assess the feasibility and safety of thoracoscopic lobectomy under spontaneous ventilation versus intubated single lung mechanical ventilation.

DETAILED DESCRIPTION:
Intubated anesthesia with single lung mechanical ventilation (SLV) is considered the standard of care in VATS. However, this type of anesthesia has been associated with several adverse effects, which can trigger complications and increase the overall surgical risk. In order to avoid intubated-anesthesia related adverse effects, spontaneous ventilation strategies have been proposed in recent years.Encouraged by the satisfactory results with a preliminary experience of spontaneous ventilated VATS, the multicentre randomized controlled clinical controled study is established to comparatively analyze the outcome of patients undergoing either nonintubated intravenous anesthesia with spontaneous ventilation (SV) or SLV VATS lobectomy, especially in safety during operation, lymph nodes resection, complication rate, muscle recovery after surgery, the difference the postoperative hospitalization time.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in clinical trials and having the ability of responsibility can be signed informed consent.
* 18-70 years old • preoperative chest CT diagnosed with "localized lung bulla" and needing surgical treatment
* Eastern Cooperative Oncology Group(ECOG) score standard ≤ 1 • ASA（American Society of Anesthesiologists score） ≤ 2
* Heart ejection fraction( EF)≥ 50

Exclusion Criteria:

* refusing to participate in clinical trials • A history of tuberculosis or other diseases could cause pleural adhesion or more pleural effusion
* BMI ≥ 25 kg/m^2
* other not suitable situation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2018-03-05 (Estimated); Primary Completion 2019-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
numbers of participants with unstable vital signs, hypoxemia or hypercapnia intraoperatively | during the surgical operation, an average of 1 hour
  the numbers of participants with unstable vital signs or hypoxemia/hypercapnia will be reported. The vital signs will be monitored through the whole surgical operation(including heart rating in beat per minute, temperature in degree Celsius, respiratory in breaths per minute and blood pressure in oxygen in millimetres of mercury ), and blood gas analysis((including partial pressure of oxygen in millimetres of mercury, partial pressure of carbon dioxide in millimetres of mercury, and so on) will be tested every 30 mins during the operation.

SECONDARY OUTCOMES:
numbers of participants with postoperative complications | from operation to discharging, an average of 1 week
  The numbers of participants with postoperative complications will be reported. The postoperative complications include postoperative respiratory complications(e.g., air leaks, lung infections, atelectasis, and bronchospasm and respiratory failure), postoperative cardiovascular complications(e.g., arrhythmias, myocardial infarction, cardiac failure) , intubated related complications(e.g., hoarseness, sore throat, and irritating cough), and other undefined complications
numbers of participants with anesthesia conversion intraoperatively in spontaneous ventilation group | during the surgical operation, an average of 1 hour
  The numbers of participants undergoing conversion from nonintubated spontaneous ventilation anaesthesia to intubated anaesthesia in nonintubated group will be reported because of hypoxemia, carbohemia, bleeding or other undefined reasons.

OTHER OUTCOMES:
the postoperative hospitalization time of every participant | through the postoperative hospitalization time, an average of 1 week
  the postoperative time point of participants meeting the discharging criteria: body T°<37.5℃, degree of blood oxygen saturation on room air>95%, no complications requiring in-hospital treatment, full lung re-expansion after chest tube removal, and white blood cell count<10×109/L

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, Ph.D, M.D., Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (2):
- China (2):
  - the First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - Fei Cui, Ph.D, M.D., Guangzhou, Guangdong

REFERENCES:
- [Background] Cui F, Liu J, Li S, Yin W, Xin X, Shao W, He J. Tubeless video-assisted thoracoscopic surgery (VATS) under non-intubated, intravenous anesthesia with spontaneous ventilation and no placement of chest tube postoperatively. J Thorac Dis. 2016 Aug;8(8):2226-32. doi: 10.21037/jtd.2016.08.02. PMID 27621880
- [Background] Peng G, Cui F, Ang KL, Zhang X, Yin W, Shao W, Dong Q, Liang L, He J. Non-intubated combined with video-assisted thoracoscopic in carinal reconstruction. J Thorac Dis. 2016 Mar;8(3):586-93. doi: 10.21037/jtd.2016.01.58. PMID 27076956
- [Background] Li S, Liu J, He J, Dong Q, Liang L, Cui F, Pan H, He J. Video-assisted transthoracic surgery resection of a tracheal mass and reconstruction of trachea under non-intubated anesthesia with spontaneous breathing. J Thorac Dis. 2016 Mar;8(3):575-85. doi: 10.21037/jtd.2016.01.62. PMID 27076955
- [Background] Liu J, Cui F, He J. Non-intubated video-assisted thoracoscopic surgery anatomical resections: a new perspective for treatment of lung cancer. Ann Transl Med. 2015 May;3(8):102. doi: 10.3978/j.issn.2305-5839.2015.04.18. PMID 26046043
- [Background] Li S, Cui F, Liu J, Xu X, Shao W, Yin W, Chen H, He J. Nonintubated uniportal video-assisted thoracoscopic surgery for primary spontaneous pneumothorax. Chin J Cancer Res. 2015 Apr;27(2):197-202. doi: 10.3978/j.issn.1000-9604.2015.03.01. PMID 25937782
- [Background] Li S, Jiang L, Ang KL, Chen H, Dong Q, Yang H, Li J, He J. New tubeless video-assisted thoracoscopic surgery for small pulmonary nodules. Eur J Cardiothorac Surg. 2017 Apr 1;51(4):689-693. doi: 10.1093/ejcts/ezw364. PMID 28007874
- [Background] Liu J, Cui F, Pompeo E, Gonzalez-Rivas D, Chen H, Yin W, Shao W, Li S, Pan H, Shen J, Hamblin L, He J. The impact of non-intubated versus intubated anaesthesia on early outcomes of video-assisted thoracoscopic anatomical resection in non-small-cell lung cancer: a propensity score matching analysis. Eur J Cardiothorac Surg. 2016 Nov;50(5):920-925. doi: 10.1093/ejcts/ezw160. Epub 2016 May 10. PMID 27165771
- [Background] Li J, Liu J, Hamblin L, Liu H, Liang L, Dong Q, He J. Simple to simplest: the tubeless technique. J Thorac Dis. 2017 Feb;9(2):222-224. doi: 10.21037/jtd.2017.02.55. No abstract available. PMID 28275463
- [Background] Dong Q, Liang L, Li Y, Liu J, Yin W, Chen H, Xu X, Shao W, He J. Anesthesia with nontracheal intubation in thoracic surgery. J Thorac Dis. 2012 Apr 1;4(2):126-30. doi: 10.3978/j.issn.2072-1439.2012.03.10. PMID 22833817
- [Background] Guo Z, Yin W, Zhang X, Xu X, Liu H, Shao W, Liu J, Chen H, He J. Primary spontaneous pneumothorax: simultaneous treatment by bilateral non-intubated videothoracoscopy. Interact Cardiovasc Thorac Surg. 2016 Aug;23(2):196-201. doi: 10.1093/icvts/ivw123. Epub 2016 May 10. PMID 27165732
- [Background] Liu J, Cui F, Li S, Chen H, Shao W, Liang L, Yin W, Lin Y, He J. Nonintubated video-assisted thoracoscopic surgery under epidural anesthesia compared with conventional anesthetic option: a randomized control study. Surg Innov. 2015 Apr;22(2):123-30. doi: 10.1177/1553350614531662. Epub 2014 May 12. PMID 24821259
- [Background] Chen JS, Cheng YJ, Hung MH, Tseng YD, Chen KC, Lee YC. Nonintubated thoracoscopic lobectomy for lung cancer. Ann Surg. 2011 Dec;254(6):1038-43. doi: 10.1097/SLA.0b013e31822ed19b. PMID 21869676